CLINICAL TRIAL: NCT02631304
Title: Delirium in Elderly Undergoing Cardiac Surgery and the Significance of CholinEsterase Activity Measured by Point of Care Method - a Prospective Observational Study
Brief Title: Delirium in Elderly Undergoing Cardiac Surgery and the Significance of CholinEsterase Activity
Acronym: DECCEP
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Ana Stevanovic, Dr. Ana Stevanovic, RWTH Aachen University
Other Study IDs: 15-162
Record Dates: First submitted 2015-12-09; First posted 2015-12-16 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Postoperative Complications
Keywords: Postoperative delirium; Cholinesterase activity; Buturylcholinesterase activity; Acetylcholinesterase activity; Elderly patients; Cardiac surgery
MeSH Terms: conditions — Postoperative Complications; Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing cardiac surgery: Elderly patients scheduled to undergo elective cardiac surgery (coronary artery bypass graft (CABG), valve surgery, combined CABG-valve surgery) with the use of cardiopulmonary bypass.
  Interventions: Procedure: Elective cardiac surgery

INTERVENTIONS:
Procedure: Elective cardiac surgery — Coronary artery bypass graft (CABG), valve surgery, combined CABG-valve surgery

SUMMARY:
The purpose of this study is to assess the association between the "point-of-care" (POC) measured ChE activity (Acetylcholinesterase (ChE) + Buturylcholinesterase (ChE)) and postoperative delirium in elderly patients undergoing cardiac surgery.

Furthermore the investigators aim to identify factors, which influence the baseline levels and the time course of ChE activity.

DETAILED DESCRIPTION:
Cardiac surgery in elderly patients is associated with serious complications, like increased morbidity, mortality and postoperative delirium with further hazardous consequences. The incidence of postoperative delirium in elderly is reported with a range from 36.6% - 54.9%. The pathophysiology of delirium is complex and the interaction of the cholinergic system and inflammation reaction is a relevant precipitant factor. It was suggested that there is a strong association between the perioperative plasma ChE activity and the inflammatory response in patients developing delirium. Patients showed a significant reduction of the total ChE activity after orthopaedic surgery, with significant lower pre- and postoperative values of AChE and BuChE and increased inflammatory response in patients developing postoperative delirium. It remains unclear if these results are applicable to other patient populations and which factors have influenced the low preoperative ChE levels. In patients suffering from a cardiac disease, a reduced total ChE respectively BuChE activity was significantly associated with mortality and long-term major adverse cardiovascular events. The investigators hypothesize that the ChE activity in peripheral blood can be used as a potential biomarker, to early detect patients at high risk for postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* ≥ 65 years of age
* Scheduled to undergo elective cardiac surgery (coronary artery bypass graft (CABG), valve surgery, combined CABG-valve surgery) with the use of CPB
* Both genders

Exclusion Criteria:

* Planned deep hypothermic arrest
* Acute / emergency procedures
* Surgery without extracorporeal circulation (ECC)
* Patients with a history of pseudocholinesterase deficiency
* Employees of the respective study centres
* Illiteracy
* Severe communication difficulties and severe vision or hearing problems
* Patients legally unable to give written informed consent
* non-fluency in German language
* Severe psychiatric or neuropsychiatric disorders
* MMSE < 24 points, short geriatric depression scale (GDS) ≥ 10 points
* Recent (<6 months) history of alcohol or drug abuse
* The participation in a drug or device trial within the previous 30 days

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Tertiary care clinic
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Acetylcholinesterase (AChE) and buturylcholinesterase (BuChE) activity | 5 days
  The perioperative AChE and BuChE activity will be assessed in the whole blood by a "point-of-care" measuring instrument (ChE check mobile ®) and the association to the incidence and duration of postoperative delirium will be determined. It will be assessed preoperative and maximum until the 5th postoperative day (POD), minimum until the 3.POD.
Delirium | 5-45 days
  Postoperative delirium will be assessed preoperative and daily with the CAM / CAM-ICU test until the 5.POD and on the discharge day from hospital. The incidence of postoperative delirium will be associated with the perioperative AChE and BuChE time course.

SECONDARY OUTCOMES:
Pre-existing patient related risk factors | 1 day
  Influence of pre-existing patient related risk factors ( demographic data, medical and surgical history assessed preoperative) on postoperative delirium and the AChE and BuChE activity.
Identification of anticholinergic concomitant medication according to the PRISCUS list | 1 day
  Number of participants with preoperative anticholinergic medication
Survey of treatment associated data | 45 days
  Survey of treatment associated data until discharge (organ dysfunctions, postoperative pain, ICU length of stay, hospital length of stay, duration of mechanical ventilation, readmission rate to ICU, operation time, surgery, anaesthesia, intraoperative and postoperative volume load, postoperative mortality, comorbidities)
Cognitive function | 45 days
  Assessment of the cognitive function preoperative and on 3.POD and at discharge,by mini mental state examination (MMSE)
Routine venous blood parameters | 5 days
  Correlation of AChE and BuChE activity and routine venous blood parameters (Hb, Platelets, Leucocytes, INR, PTT, liver-enzymes (AST, ALT, y-GT, total Bilirubin), Creatinine, BUN, Albumin, sodium and potassium) and the influence on postoperative delirium
Inflammatory markers | 5 days
  Correlation of AChE and BuChE activity to inflammatory markers in serum and the influence on postoperative delirium
Follow up measure of functional decline according to the IADL scale | 180 days
  Patients will be followed up by phone on the 30. and 180.POD. Association of AChE and BuChE activity and the functional decline on the 30. and 180.POD. The preoperative IADL scale will be compared to the data on the 30. and 180.POD to assess the functional decline
Follow up measure of mortality | 180 days
  Patients will be followed up by phone on the 30. and 180.POD. Determination of the association between the peri-operative AChE and BuChE activity and the mortality on the 30. and 180.POD
Follow up measure of the number of MACCE-events | 180 days
  Patients will be followed up by phone on the 30. and 180.POD. Association of AChE and BuChE activity and the postoperative major adverse cardiovascular and cerebral events (MACCE) on the 30. and 180.POD. The number of events will be assessed.
Health related quality of life | 180 days
  Health related quality of life measured by EuroQuol EQ-5D-5L test preoperative, on 30.POD and 180. POD
Instrumental activities of daily living | 180 days
  The Lawton Instrumental Activities of Daily Living (IADL) Scale measured preoperative, on 30.POD and 180. POD

OTHER OUTCOMES:
Gender effect on delirium assessed by CAM-ICU/CAM | 5-45 days
  Analysis of the association of postoperative delirium until 5.POD respective discharge day and the gender of the patient
Gender effects on the peri-operative AChE and BuChE activity | 5-45 days
  Measurement of the AChE and BuChE activity until 3.-5.POD. Analysis of the association of the gender of the patient and the peri-operative time-course of the AChE and BuChE activity until the 3. respective 5.POD.
Postoperative bleeding | 1 day
  Measured 12 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ana Stevanovic, MD, Principal Investigator — Department of Anesthesiology, University Hospital Aachen, Germany
Locations (1):
- Department of Anesthesiology, University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Smulter N, Lingehall HC, Gustafson Y, Olofsson B, Engstrom KG. Delirium after cardiac surgery: incidence and risk factors. Interact Cardiovasc Thorac Surg. 2013 Nov;17(5):790-6. doi: 10.1093/icvts/ivt323. Epub 2013 Jul 25. PMID 23887126
- [Background] Cerejeira J, Batista P, Nogueira V, Firmino H, Vaz-Serra A, Mukaetova-Ladinska EB. Low preoperative plasma cholinesterase activity as a risk marker of postoperative delirium in elderly patients. Age Ageing. 2011 Sep;40(5):621-6. doi: 10.1093/ageing/afr053. Epub 2011 May 15. PMID 21576115
- [Background] Rudolph JL, Inouye SK, Jones RN, Yang FM, Fong TG, Levkoff SE, Marcantonio ER. Delirium: an independent predictor of functional decline after cardiac surgery. J Am Geriatr Soc. 2010 Apr;58(4):643-9. doi: 10.1111/j.1532-5415.2010.02762.x. Epub 2010 Mar 22. PMID 20345866
- [Background] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Background] Cerejeira J, Lagarto L, Mukaetova-Ladinska EB. The immunology of delirium. Neuroimmunomodulation. 2014;21(2-3):72-8. doi: 10.1159/000356526. Epub 2014 Feb 14. PMID 24557038
- [Background] Distelmaier K, Winter MP, Rutzler K, Heinz G, Lang IM, Maurer G, Koinig H, Steinlechner B, Niessner A, Goliasch G. Serum butyrylcholinesterase predicts survival after extracorporeal membrane oxygenation after cardiovascular surgery. Crit Care. 2014 Jan 30;18(1):R24. doi: 10.1186/cc13711. PMID 24479557
- [Background] Arbel Y, Shenhar-Tsarfaty S, Waiskopf N, Finkelstein A, Halkin A, Revivo M, Berliner S, Herz I, Shapira I, Keren G, Soreq H, Banai S. Decline in serum cholinesterase activities predicts 2-year major adverse cardiac events. Mol Med. 2014 Feb 12;20(1):38-45. doi: 10.2119/molmed.2013.00139. PMID 24395570